CLINICAL TRIAL: NCT04009395
Title: Barriers and Facilitators to the Uptake of Healthy Eating Messages by Pregnant African Immigrants Living in the UK: Perspectives of Women and Midwives.
Brief Title: Barriers and Facilitators to the Uptake of Healthy Eating Messages
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Other Study IDs: V1
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Healthy Eating; Pregnancy Related

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: One-on-one in-depth interviewing
  Interventions: Other: Pregnant Women qualitative interviewing
- Midwives: One-on-one in-depth interviewing or focus group discussions
  Interventions: Other: Midwives qualitative interviewing

INTERVENTIONS:
Other: Pregnant Women qualitative interviewing — one-on-one in depth interviewing of pregnant African migrant women living in the UK on the barriers and facilitators to healthy eating in pregnancy.
  Groups: Pregnant women
Other: Midwives qualitative interviewing — one-on-one interviewing/focus group discussions with midwives on their perspectives regarding the provision of healthy eating advice to pregnant African migrant women living in the UK.
  Groups: Midwives

SUMMARY:
Obesity is on the increase and black Africans in the United Kingdom (UK) make up a significant part of this population (32%). Weight retention after pregnancy is considered as one of the leading causes of obesity. African women living in high-income countries have been found to experience more weight retention after pregnancy than Caucasian women.

Healthy eating guidelines have been provided in pregnancy in the UK (National Institute for Health and Care Excellence) and midwives have been placed to provide healthy eating advice in pregnancy, but some studies have identified that African migrants in the UK often eat and prepare food in a different way to the traditional British approach. It has also been observed that the recommended advice for pregnant women, for example, the Eat well plate and start4life are focused on traditional British foods and cooking patterns and do not include food that would be familiar to African migrants. This may impact on the meaningfulness of such guidance to African women. Therefore, this research aims to understand what prevents healthy eating or makes healthy eating easier for pregnant African migrant women in the UK. This would include understanding how healthy eating is interpreted, the cultural factors that are considered important in healthy eating, the current sources of nutrition information and midwives view on providing healthy eating advice to this population.

Eligibility

* Pregnant African migrant women (18 and above) attending ante-natal clinics in NHS hospital sites.
* Midwives who provide ante-natal advice to pregnant Africans Where Study sites will be hospitals covered by the Epsom and St Helier University trust, London North West University Healthcare National Health Service (NHS) trust and the Lewisham & Greenwich NHS trusts.

How: The study will involve one-on-one interviewing with pregnant women and midwives using hospital spaces provided by the hospital. Focus group discussions with midwives will be attempted depending on logistics. The interviews are expected to last about one hour to one and a half hours. Interview sessions will be audio-taped with the permission of the participants. Data collection is expected to last for 6 months.

DETAILED DESCRIPTION:
This study is concerned with exploring the perception of pregnant African migrant women living in the United Kingdom (UK) towards healthy eating messages and midwives perception of providing healthy eating advice to these women. The prevalence of obesity among women of reproductive age (15-49 years) including pregnant women is increasing nationally and internationally. Maternal obesity has adverse consequences for both mother and child including higher risks of perinatal mortality, Caesarean sections, preterm birth, postpartum weight retention, increased risk of macrosomia, stillbirth, congenital malformation, childhood overweight and obesity.

Currently postpartum weight retention is a significant contributor to the general obesity epidemic and obesity is a significant contributor to chronic disease burden worldwide and a public health concern. Presently, the United Kingdom (UK) has the highest level of maternal obesity in Europe with approximately 46% of women classified as either obese (20%) or overweight (26%) at their booking appointment. Non-Hispanic black women make up a significant proportion (32%) of this population. With migration rates increasing, and black Africans being considered the fastest growing ethnic group in the UK (73% of the UK population growth), the rates of obesity in the population is expected to increase. Studies have shown pre-pregnancy weight to be a significant predictor of weight changes in pregnancy and postpartum weight retention certain studies have found that more African women are overweight before pregnancy and experience more weight retention after pregnancy than Caucasian women.

However, pregnancy has been indicated as a time when public health nutrition messages can be communicated and an "opportunity for change", with women showing an inclination to modify behaviour. Therefore, globally and in the UK, there has been an increased interest in dietary/healthy eating interventions in pregnancy (sometimes in addition to physical activity) to improve folic acid intake, improve fruits and vegetables intake, limit gestational weight gain, and prevent postpartum weight retention. With systematic reviews of dietary clinical trials showing that dietary interventions in pregnancy resulted in reduction in maternal gestational weight gain and improved pregnancy outcomes. Furthermore, current clinical guidelines in the UK advocate a healthy weight before pregnancy, a healthy diet and being physically active, returning to a healthy weight post pregnancy with healthy eating guidelines provided. Midwives are also recommended and ideally placed to provide healthy eating, weight management and physical activity support to help women eat well and manage their weight during pregnancy and beyond.

Studies evaluating healthy eating adherence in pregnancy show that although a majority of pregnant women in the studies believed that their diet was healthy, just a fraction of them met the recommended dietary intake for all the food groups in pregnancy. There is very little known about the uptake of healthy eating messages/interventions and adherence to healthy eating guidelines in pregnancy amongst pregnant African migrant women living in the UK. Considering also that the healthy eating guideline is made to suit the cultural preferences of the host nation, it is imperative that dietary interventions and/or healthy eating messages targeted at this group are conducted. Following a review of literature, and discussions with practitioners, there has been no known dietary intervention in pregnancy in the UK particularly targeting pregnant migrant African women.

Evidence from systematic reviews and meta-analysis suggests that culturally adapted health interventions are effective in ethnic minority population, including those targeted at smoking cessation, physical activity and healthy diet. Health is also said to be influenced by culture-linked behaviours. Such behaviours are transmitted from elders to children and continue through generations which are evident in patterns of food selection, food preparation and mental constructions of body shape, size, functions and disease processes. Cultural adaptation involves a consideration of language, culture and context in an intervention such that it suits cultural patterns, meanings and values of the target population.The need for cultural adaptation of healthy eating messages for pregnant Africans is further buttressed by the fact that dietary behaviours of pregnant Africans post migration are not completely changed from traditional dietary practices.

Despite the need for interventions to promote healthy eating in pregnancy amongst pregnant African migrant women in the UK, very little is known about the perceptions of these women around healthy eating, factors that influence healthy eating (barriers and facilitators) and the perception of midwives regarding the provision of healthy eating advice to this population. Qualitative evidence that has considered perceptions of pregnant African women living in high income countries exist mainly in the United States and is centred on sociocultural influences regarding body size, misunderstanding about what is considered as healthy, cravings and palatability, and the belief that gaining weight indicate healthy babies.

Also qualitative studies evaluating the experiences of midwives and other healthcare providers in providing healthy eating advice to pregnant women show that although healthy eating advice was offered in pregnancy, it was not regarded as a priority. Barriers for the midwives existed in terms of topic sensitivity, inadequate training and cultural differences. Considering that qualitative evidence is context specific and might not be generalizable, it is important to explore the barriers and facilitators to healthy eating amongst pregnant African migrant women as peculiar to the United Kingdom. It is also important to explore midwives perspectives concerning the provision of healthy eating advice to this population.

This study is a formative research. Formative researches are used to determine how well an intervention would fit the needs and preferences of a group. It follows the social constructivist relativist point of view and the Medical Research Council (MRC) framework for the development and evaluation of complex interventions. The social constructivist epistemology emphasises that our reality is socially constructed based on human perception, experience, opinions, beliefs and the context of their lives and knowledge is dependent on the environment in which we live. Culture and context is emphasized with regards to understanding what occurs in the society and constructing knowledge around it. This study will attempt to understand the perception towards healthy eating by pregnant African migrant women based on their socially constructed reality within their culture and the context of living in the United Kingdom.

The MRC framework emphasizes the need to interview potential recipients of an intervention and the stakeholders with the view to identify and develop appropriate theory and increase acceptability of the intervention. Qualitative interviewing will be used to explore the concept of perceived barriers and facilitators to healthy eating during pregnancy among pregnant African migrant women living in the UK and the perception of midwives to providing healthy eating advice to pregnant African migrant women. It is hoped that evidence from this study will be used to develop a culturally adapted healthy eating intervention framework for migrant African women in the UK.

Aim To explore perceived barriers and facilitators to healthy eating amongst pregnant African migrant women in the UK and midwives perception of providing healthy eating advice to this population.

Objectives

* To determine how healthy eating is interpreted and understood by pregnant African migrant women living in the UK
* To identify the factors considered significant (barriers and facilitators) to healthy eating in this population
* To identify cultural factors considered significant to the uptake of healthy eating messages in this population
* To explore the current sources of nutrition information in pregnancy for African migrants living in the UK.
* To explore midwives perspectives on providing healthy eating advice to pregnant African migrants.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant African migrant women living in the UK (18 years and above) attending antenatal clinics in the study sites. African migrants ethnicity will be self-reported by the participants.
2. Qualified midwives working in study sites who have provided care for African migrants.

Exclusion Criteria:

1. Pregnant African migrants less than 18 years
2. Pregnant African migrants who have chronic diseases that require dietary management e.g. diabetes, hypertension, coeliac disease.
3. Adults who are unable to communicate in English or pidgin (creole spoken by sub-saharan Africans).
4. Midwives(male or female) who have not directly provided care for pregnant African migrant women will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant migrant African women(18 years and above) living in the UK will be recruited from antenatal clinics in participating NHS study sites. Also midwives who have provided care for pregnant African migrant women will be recruited also from the participating NHS study sites
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Number of pregnant women who consider healthy eating in pregnancy | 6 months
  Open ended questions will be used to gain an in depth understanding of factors considered significant to healthy eating (sources of nutrition information, barriers and facilitators) in this population.
Number of midwives who offer healthy eating advice | 6 months
  Open ended questions will be used to gain an in depth understanding of the views of mid-wives to provision of healthy eating advice to pregnant African migrants.

CONTACTS AND LOCATIONS:
Overall Officials: Aniebiet Ekong, Principal Investigator — Bournemouth University
Locations (1):
- Lewisham and Greenwich NHS Trust, Woolwich, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared when publishing results in academic journal papers and in the study protocol.
Supporting Information: Study Protocol